CLINICAL TRIAL: NCT05761171
Title: A Phase 2 Study of Revumenib (SNDX-5613) in Combination With Chemotherapy for Patients With Relapsed or Refractory KMT2A-Rearranged Infant Leukemia
Brief Title: A Study of Revumenib in Combination With Chemotherapy for Patients Diagnosed With Relapsed or Refractory Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AALL2121; NCI-2023-00503 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AALL2121 (Other: Children's Oncology Group); AALL2121 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2023-02-02; First posted 2023-03-09 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Acute Leukemia of Ambiguous Lineage; Recurrent Acute Lymphoblastic Leukemia; Recurrent Acute Myeloid Leukemia Due to Lineage Switch From Acute Leukemia of Ambiguous Lineage; Recurrent Acute Myeloid Leukemia Due to Lineage Switch From B Acute Lymphoblastic Leukemia, KMT2A-Rearranged; Recurrent Acute Myeloid Leukemia Due to Lineage Switch From Mixed Phenotype Acute Leukemia; Recurrent Mixed Phenotype Acute Leukemia; Refractory Acute Leukemia of Ambiguous Lineage; Refractory Acute Lymphoblastic Leukemia; Refractory Acute Myeloid Leukemia Due to Lineage Switch From Acute Leukemia of Ambiguous Lineage; Refractory Acute Myeloid Leukemia Due to Lineage Switch From B Acute Lymphoblastic Leukemia, KMT2A-Rearranged; Refractory Acute Myeloid Leukemia Due to Lineage Switch From Mixed Phenotype Acute Leukemia; Refractory Mixed Phenotype Acute Leukemia
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Specimen Handling; calaspargase pegol; Asparaginase; Cytarabine; fludarabine phosphate; Hydrocortisone; hydrocortisone hemisuccinate; Spinal Puncture; Methotrexate; merphos; Prednisolone; Methylprednisolone; Prednisone; deltacortene; prednylidene; revumenib; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Regimen A (revumenib, 3-drug re-induction, FLA) (Experimental): See Detailed Description.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Drug: Calaspargase Pegol; Drug: Cytarabine; Procedure: Echocardiography Test; Drug: Fludarabine Phosphate; Drug: Hydrocortisone Sodium Succinate; Procedure: Lumbar Puncture; Drug: Methotrexate; Procedure: Multigated Acquisition Scan; Drug: Prednisolone; Drug: Prednisone; Drug: Revumenib; Drug: Vincristine Sulfate
- Regimen B (revumenib, FLA) (Experimental): COMBINATION CYCLES 1-2: Patients receive revumenib PO or via NG, ND, NJ, or G-tube every 12 hours continuously, "FLA" IV on days 1-5, MTX IT, hydrocortisone IT, and cytarabine IT on day 0 and optionally on days 8, 15, and 22 of each cycle. Cycles repeat every 28 days for 2 cycles.
  MONOTHERAPY: Patients receive revumenib PO or via NG, ND, NJ, or G-tube every 12 hours continuously. Treatment repeats every 28 days for up to 12 cycles on study in the absence of disease progression or unacceptable toxicity. Patients may also receive MTX IT, hydrocortisone IT, and cytarabine IT on days 0, 8, 15 and 22 as clinically indicated.
  All patients also undergo ECHO or MUGA, collection of blood and CSF samples, lumbar puncture, and bone marrow aspiration throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Drug: Cytarabine; Procedure: Echocardiography Test; Drug: Fludarabine Phosphate; Drug: Hydrocortisone Sodium Succinate; Procedure: Lumbar Puncture; Drug: Methotrexate; Procedure: Multigated Acquisition Scan; Drug: Revumenib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and CSF samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Drug: Calaspargase Pegol — Given IV
  Other Names: Asparaginase (Escherichia coli Isoenzyme II), Conjugate with alpha-(((2,5-Dioxo-1-pyrrolidinyl)oxy)carbonyl)-omega-methoxypoly(oxy-1,2-ethanediyl); Asparlas; Calaspargase Pegol-mknl; EZN-2285; SC-PEG E. Coli L-Asparaginase; Succinimidyl Carbonate Monomethoxypolyethylene Glycol E. coli L-Asparaginase
  Arms: Regimen A (revumenib, 3-drug re-induction, FLA)
Drug: Cytarabine — Given IV and IT
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Drug: Hydrocortisone Sodium Succinate — Given IT
  Other Names: (11beta)-21-(3-Carboxy-1-oxopropyl)-11,17-dihydroxypregn-4-ene-3,20-dione, Monosodium Salt; A-Hydrocort; Buccalsone; Corlan; Cortisol Sodium Succinate; Cortop; Efcortelan; Emergent-EZ; Flebocortid; Hidroc Clora; Hycorace; Hydro-Adreson; Hydrocort; Hydrocortisone 21-Sodium Succinate; Hydrocortisone Na Succinate; Kinogen; Nordicort; Nositrol; Sinsurrene; Sodium hydrocortisone succinate; Solu-Cortef; Solu-Glyc
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap
Drug: Methotrexate — Given IT
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Procedure: Multigated Acquisition Scan — Undergo MUGA scan
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Prednisolone — Given PO or via NG, NJ, ND or G-tube
  Other Names: (11beta)-11,17,21-Trihydroxypregna-1,4-diene-3,20-dione; .delta.1-Hydrocortisone; Adnisolone; Aprednislon; Capsoid; Cortalone; Cortisolone; Dacortin H; Decaprednil; Decortin H; Delta(1)Hydrocortisone; Delta- Cortef; Delta-Cortef; Delta-Diona; Delta-F; Delta-Phoricol; Delta1-dehydro-hydrocortisone; Deltacortril; Deltahydrocortisone; Deltasolone; Deltidrosol; Dhasolone; Di-Adreson-F; Dontisolon D; Estilsona; Fisopred; Frisolona; Gupisone; Hostacortin H; Hydeltra; Hydeltrasol; Klismacort; Kuhlprednon; Lenisolone; Lepi-Cortinolo; Linola-H N; Linola-H-Fett N; Longiprednil; Metacortandralone; Meti Derm; Meticortelone; Opredsone; Panafcortelone; Precortisyl; Pred-Clysma; Predeltilone; Predni-Coelin; Predni-Helvacort; Prednicortelone; Prednisolonum; Prelone; Prenilone; Sterane
  Arms: Regimen A (revumenib, 3-drug re-induction, FLA)
Drug: Prednisone — Given PO or via NG, NJ, ND or G-tube
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
  Arms: Regimen A (revumenib, 3-drug re-induction, FLA)
Drug: Revumenib — Given PO or via NG, NJ, ND or G-tube
  Other Names: Menin-Mixed Lineage Leukemia Protein-Protein Interaction Inhibitor SNDX-5613; Menin-MLL Inhibitor SNDX-5613; Menin-MLL Interaction Inhibitor SNDX-5613; SNDX 5613; SNDX-5613; SNDX5613
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate
  Arms: Regimen A (revumenib, 3-drug re-induction, FLA)

SUMMARY:
This phase II trial tests the safety and best dose of revumenib in combination with chemotherapy, and evaluates whether this treatment improves the outcome in infants and young children who have leukemia that has come back (relapsed) or does not respond to treatment (refractory) and is associated with a KMT2A (MLL) gene rearrangement (KMT2A-R). Leukemia is a cancer of the white blood cells, where too many underdeveloped (abnormal) white blood cells, called "blasts", are found in the bone marrow, which is the soft, spongy center of the bones that produces the three major blood cells: white blood cells to fight infection; red blood cells that carry oxygen; and platelets that help blood clot and stop bleeding. The blasts crowd out the normal blood cells in the bone marrow and spread to the blood. They can also spread to the brain, spinal cord, and/or other organs of the body. The leukemia cells of some children have a genetic change in which a gene (KMT2A) is broken and combined with other genes that typically do not interact with one another; this is called "rearranged". This genetic rearrangement alters how other genes are turned on or off in the cell, turning on genes that drive the development of leukemia. Patients with KMT2A rearrangement have higher risk for cancer coming back after treatment. Revumenib is an oral medicine that directly targets the changes that occur in a cell with a KMT2A rearrangement and has been shown to specifically kill these leukemia cells in preclinical laboratory settings and in animals. Drugs used in chemotherapy, such as vincristine, prednisone, asparaginase, fludarabine and cytarabine work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. This trial is being done to find out if the combination of revumenib and chemotherapy would be safe and/or effective in treating infants and young children with relapsed or refractory KMT2A-R leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase 2 dose (RP2D) of revumenib administered in combination with chemotherapy in patients with relapsed or refractory (R/R) KMT2A-rearranged (KMT2A-R) acute lymphoblastic leukemia (ALL).

II. To estimate the minimal residual disease (MRD) negative remission rate of patients with R/R infant KMT2A-R ALL treated with revumenib in combination with chemotherapy.

SECONDARY OBJECTIVES:

I. To characterize the pharmacokinetics (PK) of revumenib administered with chemotherapy in patients with R/R infant KMT2A-R ALL.

II. To estimate the 18-month event-free survival (EFS) of patients with R/R infant KMT2A-R ALL treated with revumenib in combination with chemotherapy.

III. To estimate 18-month overall survival (OS) of patients with R/R infant KMT2A-R ALL treated with revumenib in combination with chemotherapy.

IV. To characterize the tolerability of revumenib given as monotherapy in patients with R/R infant KMT2A-R ALL.

EXPLORATORY OBJECTIVE:

I. To assess the biologic activity of revumenib administered with chemotherapy in patients with R/R KMT2A-R ALL.

II. To estimate the MRD negative remission rate of patients with R/R non-infant KMT2A-R ALL treated with revumenib in combination with chemotherapy.

III. To characterize the PK of calaspargase pegol-mknl and describe associated toxicities for patients with R/R KMT2A-R ALL.

IV. To describe the anti-cancer therapies received before and after administration of revumenib by patients with R/R KMT2A-R ALL.

OUTLINE: Patients with acute lymphoblastic leukemia (ALL), acute leukemia of ambiguous lineage (ALAL), or mixed phenotype acute leukemia (MPAL) are assigned to 1 of 2 regimens, by physician discretion. Patients with acute myeloid leukemia (AML) are assigned to Regimen B.

REGIMEN A:

COMBINATION CYCLE 1: Patients receive revumenib orally (PO) or via nasogastric (NG), nasojejunal (NJ), nasoduodenal (ND) or gastrostomy tube (G-tube) every 12 hours continuously. Patients also receive "3-drug re-induction" consisting of vincristine intravenously (IV) on days 1, 8, 15, and 22, prednisone or prednisolone PO or via NG, ND, NJ, or G-tube twice daily (BID) on days 1-28, calaspargase pegol-mknl IV over 1-2 hours on day 4, as well as methotrexate (MTX) intrathecally (IT) on days 1 and 8 then optionally weekly, hydrocortisone IT, and cytarabine IT. Patients who have early progressive disease may continue to Combination Cycle 2 early before fully completing cycle 1.

COMBINATION CYCLE 2: Patients receive revumenib PO or via NG, NJ, ND, or G-tube every 12 hours continuously, "FLA" consisting of fludarabine IV over 60 minutes and high-dose cytarabine IV over 1-3 hours on days 1-5. After completion of Combination Cycle 2, patients who experienced early progressive disease in Combination Cycle 1 continue to Combination Cycle 3. All other patients proceed to Monotherapy.

COMBINATION CYCLE 3: Patients receive revumenib PO or via NG, NJ, ND, or G-tube every 12 hours continuously, "FLA" as in Combination Cycle 2, MTX IT, hydrocortisone IT, and cytarabine IT on day 0.

MONOTHERAPY: Patients receive revumenib PO or via NG, NJ, ND, or G-tube every 12 hours continuously. Patients may also receive MTX IT, hydrocortisone IT, and cytarabine IT as clinically indicated.

REGIMEN B:

COMBINATION CYCLES 1-2: Patients receive revumenib PO or via NG, ND, NJ, or G-tube every 12 hours continuously, "FLA" IV on days 1-5, MTX IT, hydrocortisone IT, and cytarabine IT on day 0 and optionally on days 8, 15, and 22 of each cycle. Cycles repeat every 28 days for 2 cycles.

MONOTHERAPY: Patients receive revumenib PO or via NG, ND, NJ, or G-tube every 12 hours continuously. Treatment repeats every 28 days for up to 12 cycles on study in the absence of disease progression or unacceptable toxicity. Patients may also receive MTX IT, hydrocortisone IT, and cytarabine IT on days 0, 8, 15 and 22 as clinically indicated.

All patients also undergo echocardiography (ECHO) or multigated acquisition scan (MUGA), collection of blood and cerebrospinal fluid (CSF) samples, lumbar puncture, and bone marrow aspiration throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 1 month to < 6 years old at the time of study enrollment and must have had initial diagnosis of leukemia at < 2 years old.
* Patients must have KMT2A-rearranged acute lymphoblastic leukemia (ALL), acute leukemia of ambiguous lineage (ALAL), or mixed phenotype acute leukemia (MPAL), which is determined to be refractory or in first marrow relapse. All patients must undergo cytogenetics and fluorescence in situ hybridization (FISH) testing of a relapsed/refractory blast sample at a Children's Oncology Group (COG)-approved laboratory for KMT2A-R status determination and the presence of a KMT2A- rearrangement must be confirmed by central review. Cytogenetics results must be submitted for central review by Day 10 of protocol therapy, for confirmation of KMT2A-R status. Patients enrolled with refractory disease may utilize initial diagnostic cytogenetics for eligibility and submission for central review if testing was performed at a COG approved laboratory. Patients will be eligible to remain on protocol therapy if KMT2A-R is confirmed by central review. Additional methods of assessing for KMT2A-R may be considered if FISH does not detect the rearrangement.
* Disease status at time of enrollment must be one of the following:

  * First relapse (untreated): Any recurrence of marrow disease, with or without other extramedullary sites(s), at any point after achieving remission ("remission-1", per definition below) and meeting one of the below criteria. Patients must not have received any disease-directed therapy for the marrow relapse prior to enrollment, other than permitted cytoreduction.

    * Relapse M1: M1 morphology (< 5% blasts) + at least 2 confirmatory tests showing >= 1% blasts (testing includes flow, cytogenetics, polymerase chain reaction [PCR]/next-generation sequencing [NGS] of immunoglobulin [Ig]/T-cell receptor [TCR] rearrangement, and/or PCR or NGS of fusion gene identical to diagnosis), OR
    * Relapse M2: M2 morphology (5-25% blasts) + 1 confirmatory test showing > 1% blasts, OR
    * Relapse M3: M3 morphology (> 25% blasts)
  * Primary refractory, or failure to achieve remission-1: remission-1 is defined as < 1% marrow blasts by flow MRD and resolution of extramedullary disease following at least 2 courses of frontline chemotherapy. Patients who receive 2 courses of chemotherapy and 1 course of blinatumomab are also eligible, but no further treatment attempts beyond that are permitted
* Central nervous system (CNS) disease: Patients must have CNS1 or CNS2 status and no clinical signs or neurologic symptoms suggestive of CNS leukemia, such as cranial palsy.

  * Patients with CNS3 disease may receive antecedent intrathecal chemotherapy to achieve CNS1 or CNS2 status prior to enrollment.
  * Patients with a history of CNS chloromatous disease are required to have no radiographic evidence of CNS disease prior to enrollment.
* White blood cell (WBC) must be < 50,000/uL at the time of study enrollment. Patients can receive cytoreduction with hydroxyurea and/or corticosteroids for up to 7 days prior to enrollment.
* Patients >= 12 months of age must have a performance status by Lansky Scale of >= 50%.
* Patients must be able to take enteral medications. Acceptable routes of administration for revumenib (SNDX-5613) include: oral (PO), nasogastric (NG) tube, nasojejunal (NJ) tube, nasoduodenal (ND), and gastrostomy tube (G-tube).
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study

  * Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive:

    * >= 14 days must have elapsed after the completion of other cytotoxic therapy, including patients who relapse during pre-Maintenance upfront therapy, with these specific exceptions: cytoreduction with hydroxyurea and/or corticosteroids, and intrathecal chemotherapy, which have no required washout periods. For patients who relapse during upfront Maintenance therapy, >= 7 days must have elapsed after the last dose of chemotherapy. Additionally, patients must have fully recovered from all acute toxic effects of prior therapy.

      * NOTE: Cytoreduction with hydroxyurea and/or corticosteroids is permitted prior to enrollment for patients with WBC >= 50,000/uL, and by provider discretion regardless of WBC, to reduce potential risk of differentiation syndrome with revumenib initiation. Hydroxyurea and/or corticosteroids may be given for up to 7 days, with no wash-out required.
      * NOTE: No waiting period is required for patients having received intrathecal cytarabine, methotrexate, and/or hydrocortisone. Intrathecal chemotherapy that is given up to 7 days prior to the initiation of protocol therapy counts as protocol therapy and not prior anti-cancer therapy. Intrathecal chemotherapy given > 7 days prior does not count as protocol therapy.
      * NOTE: Prior exposure to fludarabine and cytarabine (FLA) is permitted.
  * Anti-cancer agents not known to be myelosuppressive (e.g., not associated with reduced platelet or absolute neutrophil count [ANC] counts): >= 7 days after the last dose of agent.
  * Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1. There is an exception for blinatumomab infusions, for which patients must have been off for at least 3 days and all drug related toxicity must have resolved to grade 2 or lower as outlined in the inclusion/exclusion criteria.
  * Hematopoietic growth factors: >= 14 days after the last dose of a long-acting growth factor (e.g., pegfilgrastim) or >= 7 days for short-acting growth factor. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair and the study-assigned Research Coordinator.
  * Interleukins, interferons and cytokines (other than hematopoietic growth factors): >= 21 days after the completion of interleukins, interferon, or cytokines
  * Stem cell infusions (with or without total body irradiation (TBI):

    * Allogeneic (non-autologous) bone marrow or stem cell transplant, or stem cell boost: >= 84 days after infusion
    * Donor leukocyte infusion: >= 28 days
  * Cellular therapy: >= 28 days after the completion of any type of cellular therapy (e.g., modified T cells, natural killer [NK] cells, dendritic cells, etc.)
  * Radiation therapy (XRT)/external beam irradiation including protons: >= 14 days after local XRT; >= 84 days after TBI, craniospinal XRT or if radiation to >= 50% of the pelvis; >= 42 days if other substantial bone marrow radiation.
* A creatinine based on age as follows:

  * Age 1 month to < 6 months: maximum creatinine 0.4 mg/dL
  * Age 6 months to < 1 year: maximum creatinine 0.5 mg/dL
  * Age 1 to < 2 years: maximum creatinine 0.6 mg/dL
  * Age 2 to < 6 years: maximum creatinine 0.8 mg/dL OR

    * a 24-hour urine creatinine clearance >= 70 mL/min/1.73 m^2 OR
    * a glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2. GFR must be performed using direct measurement with a nuclear blood sampling method OR direct small molecule clearance method (iothalamate or other molecule per institutional standard).
  * NOTE: Estimated GFR (eGFR) from creatinine, cystatin C or other estimates are not acceptable for determining eligibility.
* A direct bilirubin =< 1.5 x upper limit of normal (ULN) for age, unless disease related
* Serum glutamic-pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L (3 x ULN) unless disease related.

  * Note: For the purpose of eligibility, the ULN for SGPT (ALT) has been set to the value of 45 U/L
* Shortening fraction of >= 27% by echocardiogram, or ejection fraction of >= 50% by radionuclide angiogram.
* Corrected QT interval using Fridericia formula (QTcF) of < 450 msec (using the average of triplicate measurements)
* NOTE: There are no specific electrolyte parameters for eligibility. However, it should be noted that, to limit QTc prolongation risk, patients must maintain adequate potassium and magnesium levels to initiate and continue revumenib (SNDX-5613) on protocol therapy.
* Patients must be able to comply with the safety monitoring requirements of the study, in the opinion of the treating investigator.

Exclusion Criteria:

* Patients with isolated extramedullary leukemia.
* Patients diagnosed with Down syndrome.
* Patients known to have one of the following syndromes:

  * Bloom syndrome, ataxia-telangiectasia, Fanconi anemia, Kostmann syndrome, Shwachman syndrome, or any other known bone marrow failure syndrome.
* Patients with a secondary KMT2A-R leukemia that developed after treatment of prior malignancy with cytotoxic chemotherapy.
* Patients with a history of congenital prolonged QT syndrome, congestive heart failure or uncontrolled arrhythmia in the past 6 months prior to study enrollment.
* Patients with an active, uncontrolled infection, further defined below:

  * Positive bacterial blood culture within 48 hours of study enrollment
  * Fever above 38.2 degrees Celsius (C) within 48 hours of study enrollment with clinical signs of infection. Fever that is determined to be due to tumor burden is allowed if patients have documented negative blood cultures for at least 48 hours prior to enrollment and no concurrent signs or symptoms of active infection or hemodynamic instability
  * A positive fungal culture within 30 days of study enrollment or active therapy for presumed invasive fungal infection
  * Patients may be receiving IV or oral antibiotics to complete a course of therapy for a prior documented infection as long as cultures have been negative for at least 48 hours and signs or symptoms of active infection have resolved. For patients with Clostridium (C.) difficile diarrhea, at least 72 hours of antibacterial therapy must have elapsed and stools must have normalized to baseline
  * Active viral or protozoal infection requiring IV treatment
  * Human immunodeficiency virus (HIV)-infected patients are eligible if on effective anti-retroviral therapy that does not interact with planned study agents and with undetectable viral load within 6 months of enrollment.
* Patients with active acute graft-versus-host disease (GVHD) > grade 0 (unless skin only), or chronic GVHD > mild (unless skin only) are not eligible. Patients with acute or chronic skin GVHD that is =< grade 1, or chronic skin GVHD that is graded as mild are eligible.
* Patients who have received a prior solid organ transplantation.
* Patients with known Charcot-Marie-Tooth disease, if treating on Regimen A (with vincristine).
* CYP3A4 Inhibitors or Inducers: Patients who require concomitant therapy with strong CYP3A4 inhibitors or moderate or strong CYP3A4 inducers, as these are prohibited during the chemotherapy combination cycles. These agents should be discontinued at least 5 half-lives prior to starting protocol therapy. Concomitant use of strong CYP3A4 inhibitor -azole antifungals are permitted during the revumenib (SNDX-5613) monotherapy cycles, with appropriate revumenib (SNDX-5613) dose modification
* P-glycoprotein (P-gp) inhibitors or inducers: Vincristine is a substrate for P-gp. Concomitant use of P-gp inhibitors or inducers with vincristine (patients receiving Regimen A Cycle 1) should be avoided.
* Investigational drugs: Patients who are currently receiving another investigational drug.
* Anti-cancer agents: Patients who are currently receiving other anti-cancer agents (exceptions: hydroxyurea and corticosteroids, which may be used as cytoreduction prior to enrollment).
* Anti-GVHD agents: Patients who are receiving cyclosporine, tacrolimus, or other systemic agents to treat graft-versus-host disease post bone marrow transplant. Patients should discontinue anti-GVHD agents > 7 days prior to enrollment and have no evidence of worsening GVHD. Topical steroids are permitted.
* Patients who have previously been treated with revumenib (SNDX-5613). Prior exposure to other menin inhibitors is permitted.
* All patients and/or their parents or legal guardians must sign a written informed consent.
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met.

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) for lymphoid directed chemotherapy block (Safety Phase) | At the end of Cycle 1 of Regimen A (each cycle is a minimum of 29 days)
  Regimen A Cycle 1 will be used for determination of recommended phase 2 dose (RP2D)-lymphoid (L) directed chemotherapy block. A patient will be considered as being evaluable for DLT if: (1) the patient receives at least 66 doses of the first planned 28 days (84 doses) of revumenib for the cycle (for patients with delayed revumenib shipment, will count 28 days from the start of revumenib); or (2) the patient experiences a DLT after the start of revumenib in Cycle 1.
Incidence of dose-limiting toxicities (DLTs) for myeloid directed chemotherapy block (Safety Phase) | At the end of Cycle 1 of Regimen B and at the end of Cycle 2 of Regimen A (each cycle is a minimum of 29 days)
  Regimen B Cycle 1 and Regimen A Cycle 2 will be used for determination of RP2D-myeloid (M) directed chemotherapy block. For each cycle mentioned above, a patient will be considered as being evaluable for DLT if: (1) the patient receives at least 66 doses of the first planned 28 days (84 doses) of revumenib for the cycle (for patients with delayed revumenib shipment, will count 28 days from the start of revumenib); or (2) the patient experiences a DLT after the start of revumenib in that cycle. For determination of RP2D-M, patients in Regimen A who have experienced a DLT in Cycle 1 or who have been evaluated as having Early Progressive Disease in Cycle 1 are excluded.
Minimal residual disease (MRD) negative remission rate in patients with relapsed/refractory (R/R) infant KMT2A-R ALL (Expansion Phase) | Up to 3 cycles of combination therapy (each cycle is a minimum of 29 days)
  A patient with R/R infant KMT2A-R ALL will be included in the primary analysis of MRD negative remission rate if the patient is enrolled at RP2D-L and RP2D-M (in the safety phase or the expansion phase) and receives at least one dose of protocol treatment. This response rate will be estimated using the approach of Jung and Kim. The corresponding 95% confidence interval will be calculated using the approach of Koyama and Chen.

SECONDARY OUTCOMES:
Proportion of patients achieving desired SNDX-5613 pharmacokinetics (PK) during the expansion phase | Up to 2 years from enrollment
  Analyses will be conducted for lymphoid and myeloid blocks separately and then combined. Will monitor if there is evidence that the proportion of patients achieving desired PK is considerably lower than 90% using the Pocock stopping boundaries.
Estimation of 18-month event-free survival (EFS) rate in patients with R/R infant KMT2A-R ALL | Time from date of enrollment to date of treatment failure, relapse, second or secondary malignancy (SMN), or death due to any cause, whichever occurs first, assessed up to 18 months
  Will be estimated using the Kaplan-Meier method.
Estimation of 18-month overall survival (OS) rate in patients with R/R infant KMT2A-R ALL | Time from date of enrollment to death due to any cause, assessed up to 18 months
  Will be estimated using the Kaplan-Meier method.
Characterization of tolerability of revumenib given as monotherapy in patients with R/R infant KMT2A-R ALL | Up to 2 years from enrollment
  Grade 3+ adverse events (AEs) will be summarized among patients receiving monotherapy, by cycles, and the proportion of patients having grade 3+ AEs will be estimated.

OTHER OUTCOMES:
Changes in KMT2A-R transcriptional program | Up to 5 years from enrollment
  Ribonucleic acid (RNA) will be isolated from cryopreserved leukemic cell suspensions and exploratory analysis of RNA sequencing (Seq) will be performed. Principal component analysis and gene set enrichments will be used to compare overall transcriptional signatures, and specifically the reported KMT2A-R dependent gene sets, comparing paired pre-treatment and post-treatment samples. Correlations between changes in RNA-Seq and patient's clinical response to SNDX-5613 as well as pharmacokinetic parameters and menin displacement will be described.
Changes to menin displacement | Up to 5 years from enrollment
  Pre-treatment and post-treatment paired samples will be tested for menin occupancy by CUT&RUN, and changes to informative histone modifications/protein complexes evaluated by CUT&Tag. The degree of reduction in menin binding to specific target genes will be correlated with clinical response and pharmacokinetic parameters, as well as biologic transcriptional changes.
MRD negative remission rates in patients with R/R non-infant KMT2A-R ALL | Up to 3 cycles of combination therapy (each cycle is a minimum of 29 days)
  MRD negative remission rates will be summarized.
PK of calaspargase pegol-mknl and the associated toxicities for patients with R/R KMT2A-R ALL | Up to 5 years from enrollment
  Analyses will be conducted for lymphoid and myeloid blocks separately and then combined and will be restricted to patients who receive calaspargase-pegol-mknl. These analyses will be exploratory and descriptive.
Anti-cancer therapies received before and after administration of revumenib by patients with R/R KMT2A-R ALL | Up to 5 years from enrollment
  The types of anti-cancer therapies received by patients before or after administration of revumenib will be described. The association between the anti-cancer therapies patients received prior to enrollment and response may also be assessed. The association between the anti-cancer therapies received after revumenib and EFS or OS may be assessed. These analyses will be exploratory and descriptive.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly E Faulk, Principal Investigator — Children's Oncology Group
Locations (84):
- United States (75):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- Canada (9):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec